CLINICAL TRIAL: NCT06740240
Title: 68Ga-FAPI-Biotin PET/CT in Patients With Various Types of Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-FAPI-Biotin
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-FAPI-Biotin PET/ CT (Experimental): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI-Biotin. Tracer of 68Ga-FAPI-Biotin will be used to detect tumors by PET/CT.
  Interventions: Drug: 68Ga-FAPI-Biotin
- 68Ga-FAPI/18F-FDG PET/CT (Active Comparator): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI or 3.7 MBq (0.1 mCi)/Kg18F-FDG. Tracer of 68Ga-FAPI/18F-FDG will be used to detect tumors by PET/CT.
  Interventions: Drug: 68Ga-FAPI/18F-FDG

INTERVENTIONS:
Drug: 68Ga-FAPI-Biotin — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI-Biotin. Tracer doses of 68Ga-FAPI-Biotin will be used to detect tumors by PET/CT
  Arms: 68Ga-FAPI-Biotin PET/ CT
Drug: 68Ga-FAPI/18F-FDG — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-FAPI or 3.7 MBq (0.1 mCi)/Kg 18F-FDG. Tracer doses of 68Ga-FAPI/18F-FDG will be used to detect tumors by PET/CT.
  Arms: 68Ga-FAPI/18F-FDG PET/CT

SUMMARY:
As a new dual targeting PET radiotracer, 68Ga-FAPI-Biotin is promising as an excellent imaging agent applicable to various cancers. In this study, we observed the safety, biodistribution and radiation dosimetry of 68Ga-FAPI-Biotin in patients with various types of cancer and compared them with the results of 68Ga-FAPI or 18F-FDG imaging to evaluate the dosimetric characteristics and diagnostic efficacy of 68Ga-FAPI.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is highly expressed in the stroma of a variety of human cancers and is therefore considered promising for guiding targeted therapy. The recent development of quinoline-based PET tracers that act as FAP inhibitors (FAPIs) demonstrated promising results preclinically and already in a few clinical cases. Biotin is overexpressed in various tumor cells and underexpressed in normal cells. We assume that expanding molecular probes targeting FAPI and biotin with dual targets to enhance the targeting ability of the tracer, improve the sensitivity and specificity of tumor lesion detection. 68Ga-FAPI-Biotin is a novel dual targeting tracer. The present study aimed to evaluate the biodistribution, pharmacokinetics, and dosimetry of 68Ga-FAPI-Biotin, and performed a head-to-head comparison with 68Ga-FAPI or 18F-FDG PET/CT scans in patients with various cancers.

ELIGIBILITY:
Inclusion Criteria:

Various solid tumors with available histopathological findings; Signed informed consent.

Exclusion Criteria:

Pregnant or lactational women; who suffered from severe hepatic and renal insufficiency.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 3 months.
  Sensitivity and Specificity of 68Ga-FAPI-Biotin in Patients With Various Types of Cancer and compare it with 68Ga-FAPI/18F-FDG PET/CT.

SECONDARY OUTCOMES:
SUV of tumors | through study completion, an average of 3 months.
  Compare the SUV of tumors between 68Ga-FAPI-Biotin PET/CT and 68Ga-FAPI/18F-FDG PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, China